CLINICAL TRIAL: NCT01857713
Title: A Multi-Center, Non-Randomized, Prospective Study of the Reza Band™ Upper Esophageal Sphincter (UES) Assist Device for the Treatment of Esophagopharyngeal Reflux
Brief Title: Treatment of Extraesophageal Reflux With the Reza Band UES Assist Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somna Therapeutics, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RB-001-02
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-05

CONDITIONS: Laryngopharyngeal Reflux
MeSH Terms: conditions — Laryngopharyngeal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reza Band UES Assist Device (Active Comparator): Patient is own control. Compare baseline to last follow-up after using device
  Interventions: Device: Reza Band UES Assist Device

INTERVENTIONS:
Device: Reza Band UES Assist Device — Device is worn by patient to reduce or eliminate laryngopharyngeal reflux

SUMMARY:
The purpose of the study is to determine the safety and effectiveness of non-invasive Reza Band UES Assist Device for the treatment of esophagopharyngeal reflux with extra-esophageal symptoms (chronic cough, choking, aspiration, chronic post nasal drip, globus, sore throat, throat clearing).

DETAILED DESCRIPTION:
The purpose of the study is to determine the safety and effectiveness of non-invasive Reza Band UES Assist Device for the treatment of esophagopharyngeal reflux with extra-esophageal symptoms (chronic cough, choking, aspiration, chronic post nasal drip, globus, sore throat, throat clearing). Reza Band is to be worn when sleeping. The patient will put the Reza Band on at bedtime and take it off upon waking.

This is a prospective, non-randomized, open label, multicenter study designed to assess the safety and effectiveness of the Reza Band. At up to 5 investigational sites, up to 100 subjects will be enrolled.

The primary effectiveness endpoint is to be evaluated by the Reflux Symptom Index (RSI). Success is defined as >25% reduction in the RSI at the last follow-up, as compared to the baseline RSI. The RSI is a validated nine-item patient-administered outcome questionnaire designed to document symptoms and severity. Patients are asked to rate how nine problems have affected them on a scale of 0 (no problem) to 5 (severe problem), with a maximum total score of 45.

All adverse reactions being reported will be evaluated with the frequency and percent of subjects of each reaction being summarized by severity and by relationship to the Reza Band. Since some subjects may report the same event several times (e.g., redness), the first occurrence of the worst reported case of the event will be used for the purpose of analysis.

The incidence of site reactions, including laryngospasm, choking, pain, cough and hoarseness will be summarized. Exact 95% confidence intervals for the incidence rate of site reactions will be presented.

ELIGIBILITY:
Inclusion Criteria:

* 18 year of age or older
* The patient must be willing and able to provide informed consent.
* Understands the clinical study requirements and is able to comply with follow-up schedule.
* Clinically diagnosed with esophagopharyngeal reflux with extra-esophageal symptoms (i.e., chronic cough, choking, aspiration, chronic post nasal drip, globus, sore throat, throat clearing)
* Reflux Symptom Index (RSI) >13

Exclusion Criteria:

* Currently being treated with another investigational medical device and/or drug
* Currently receiving treatment for sleep apnea with continuous positive airway pressure (CPAP)
* The patient is female and is of child bearing potential and is not using an acceptable method of birth control, or is pregnant or breast feeding.
* Previous head or neck surgery or radiation
* Carotid artery disease, thyroid disease, or history of cerebral vascular disease
* Suspected esophageal cancer
* Has either a pacemaker or implanted cardioverter defibrillator (ICD)
* Nasopharyngeal cancer
* Previously undergone Nissen Fundoplication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Dr. Alan Raymond, New York, New York
  - Madison ENT & Facial Plastic surgery, New York, New York
  - Vanderbilt University, Nashville, Tennessee
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
  - Aurora Health Care, Summit, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Fitted With Reza Band UES Assist Device: Patients were fitted with the Reza Band UES Assist Device and served as their own control. Baseline measures were comported to follow-up visit measures.
Period: Overall Study
Arm/Group | Fitted With Reza Band UES Assist Device
Started | 95
Completed | 89
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: Patients who enrolled in the study and had a Reza Band fitted by the Investigator and who had at least one post-baseline RSI assessment were included.
Groups:
- Fitted With Reza Band UES Assist Device: Patients were their own control and Fitted with Reza Band UES Assist Device. Results were obtained by measuring symptoms at baseline and then compared at each of the prescribed follow-up visits.
Arm/Group | Fitted With Reza Band UES Assist Device
Number analyzed (Participants) | 95
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.8 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 29
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 4
  Caucasian | 77
  Hispanic | 8
  Asian | 1
  Other | 1
  Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 95
Weight [Mean (Standard Deviation); unit: pounds] | 160.0 (31.3)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.5 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the Reflux Symptom Index (RSI) at 4 Weeks
Description: The RSI is a validated nine-item patient-administered outcome questionnaire designed to document symptoms and severity. Patients are asked to rate how nine problems have affected them on a scale of 0 (no problem) to 5 (severe problem), with a maximum total score of 45).
Time Frame: 4 Weeks minus Baseline
Measure: Mean (Standard Deviation); unit: Per Cent Change
Groups:
- Reza Band: Participants fitted with Reza Band UES Assist Device
Arm/Group | Reza Band
Number analyzed (Participants) | 89
Per Cent Change | -54.3 (27.1)
Statistical Analysis 1: Comparison: Reza Band; The sample size was based on the primary effectiveness variable (% reduction in RSI from Baseline to Week 4). It was assumed that the study would be successful if the mean % reduction is significantly greater than 25%. Assuming a 35% reduction in RSI, a power of 80%, one-sided significance level of 0.05, 85 subjects are required for the study. It was decided to recruit up to 100 subjects for this study; Test type: Non-Inferiority or Equivalence — It was assumed that the study would be successful if the mean % reduction is significantly greater than 25%. Assuming a 35% reduction in RSI, a power of 80%, one-sided significance level of 0.05, 85 subjects are required for the study. It was decided to recruit up to 100 subjects for this study; p < 0.05, t-test, 1 sided

2. Primary Outcome: Primary Safety
Description: Adverse reactions reported were evaluated with the frequency and percent of subjects of each reaction being summarized by severity and by relationship to the Reza Band UES Assist Device.
Time Frame: 4 Week Follow-up
Population: Patients that have been clinically diagnosed with esophagopharyngeal reflux with extra-esophageal symptoms (i.e., chronic cough, choking, aspiration, chronic post nasal drip, globus, sore throat, throat clearing).
Measure: Number; unit: % Reporting Any Adverse Event
Groups:
- Fitted With Reza Band UES Assist Device: Patients that have been clinically diagnosed with esophagopharyngeal reflux with extra-esophageal symptoms (i.e., chronic cough, choking, aspiration, chronic post nasal drip, globus, sore throat, throat clearing).
Arm/Group | Fitted With Reza Band UES Assist Device
Number analyzed (Participants) | 95
% Reporting Any Adverse Event | 58.6

3. Secondary Outcome: SF-36 Short Form Health Survey - 4 Week Follow-up Score Compared to Baseline Score
Description: The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: 4 Weeks minus Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in Units on a Scale
Arm/Group | Fitted With Reza Band UES Assist Device
Number analyzed (Participants) | 89
Change in Units on a Scale | 0.56 (6.88)

4. Secondary Outcome: Functional Outcomes of Sleep Questionnaire (FOSQ)
Description: The FOSQ is a self-report measure (0-4 for each of 30 questions) designed to assess the impact of disorders of excessive sleepiness (DOES) on multiple activities of everyday living that includes areas of physical, mental and social functioning. Scores can range from 0 (worst possible outcome) to 120 (best possible outcome). Zero (0) is defined as not doing that specific activity for other reasons.
Time Frame: 4 Weeks minus Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in Units on a Scale
Groups:
- Fitted With Reza Band UES Assist Device: Patients were fitted with the Reza Band UES Assist Device and Patients that have been clinically diagnosed with esophagopharyngeal reflux with extra-esophageal symptoms (i.e., chronic cough, choking, aspiration, chronic post nasal drip, globus, sore throat, throat clearing).
Arm/Group | Fitted With Reza Band UES Assist Device
Number analyzed (Participants) | 89
Change in Units on a Scale | 0.80 (11.04)

5. Other Pre Specified Outcome: Patient Satisfaction
Description: Patients provide their perception of the device at the end of the study.
Time Frame: 4 Weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Investigator Questionnaire
Description: Investigators provide their perception of the device at the end of the study.
Time Frame: 4 Weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from patient diaries as well as at the time of follow-up visits by the investigators. The events were noted throughout the length of the study, 4 weeks from the initial fitting of the Reza Band
Groups:
- Fitted With Reza Band UES Assist Device: Patients were fitted with the Reza Band UES Assist Device and were their own controls. Baseline measures were compared to each of the prescribed follow-up visit measures.
Arm/Group | Fitted With Reza Band UES Assist Device
Serious Adverse Events (participants affected / at risk) | 0/95
Other Adverse Events (participants affected / at risk) | 7/95
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fitted With Reza Band UES Assist Device (N=95)
Reza Band Comfort (Social circumstances) | 1 — Woke up because Reza Band was too uncomfortable
Post Nasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 — Patient reported post nasal drip while wearing Reza Band
Temporomandibular Joint Disorders (General disorders) | 1 — TMJ was noted following a dental procedure. Determined by the investigator to not be related to the device.
Bruised neck (Musculoskeletal and connective tissue disorders) | 1 — Patient reported sleeping on stomach which resulted in bruising of the neck from the device.
Biopsies due to Colonoscopy (Gastrointestinal disorders) | 1 — Two biopsies taken as a result of colonoscopy. Determined by the investigator not to be related to the device.
Fell Down (General disorders) | 1 — Fell down in garage and injured foot. Determined by the investigator not to be related to the device.
Throat infection (Ear and labyrinth disorders) | 1 — Infection that was ongoing and treated by the investigator with antibiotics. Determined by the investigator not to be related to the device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No